CLINICAL TRIAL: NCT00934310
Title: Patient Safety: Introduction of the Surgical Safety Checklist and Patient Outcome Assessment in an Academic Ambulatory Hospital
Brief Title: Introduction of the Surgical Safety Checklist
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Women's College Hospital (Other); Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Pamela J. Morgan, Dr. Pamela J Morgan, Women's College Hospital
Other Study IDs: 2009-0017-E
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Postoperative Complications
Keywords: Patient Safety; Team work; Communication; Ambulatory surgical patients
MeSH Terms: conditions — Postoperative Complications; Communication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ambulatory Surgical Patients 1: The nature of the operating room "time out" for ambulatory surgical patients will be examined before implementation of the World Health Organization's Surgical Safety Checklist.
- Ambulatory Surgical Patients 2: The nature of the operating room "time out" for ambulatory surgical patients will be examined after implementation of the World Health Organization's Surgical Safety Checklist.Ambulatory surgical patients

SUMMARY:
In January of 2007, the World Health Organization's (WHO) World Alliance for Patient Safety initiated a project called "Safe Surgery Saves Lives" to identify minimum standards of surgical care that can be universally applied across countries and settings. Through a two year process involving international input from surgeons, anesthesiologists, nurses, infectious disease specialists, epidemiologists and others, the WHO created a surgical safety checklist that encompasses a simple set of surgical safety standards that can be used in any surgical setting. Each safety step on the checklist is simple, widely applicable, and measurable. The Surgical Safety Checklist was piloted in 8 hospitals around the world and results demonstrated a significant decrease in death rate and postoperative complications.

This study proposes to introduce an adaptation of the Surgical Safety Checklist for an ambulatory care surgical program and to assess the efficacy of its adaptation and implementation on staff safety attitudes and patient outcomes. Specific ambulatory-based items will be included in the checklist and patient outcomes will be assessed using the Institute for Health Improvement's Perioperative Surgical Outcomes Tool which will also be adapted for use for the ambulatory setting as well as routine follow up phone calls with patients on the 1st postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory surgical patient

Exclusion Criteria:

* in-patient or any patient who is planning to be admitted to hospital postoperatively

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ambulatory surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The primary outcomes of this study are to determine if there are significant differences in (a) staff safety attitudes and (b) incidence of postoperative complications before and after implementation of the Surgical Safety Checklist | Before and after implementation of checklist
The primary outcomes of this study are to determine if there are significant differences in (a) staff safety attitudes and (b) incidence of postoperative complications before and after implementation of the Surgical Safety Checklist | Before and after implementation of the safety checklist

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J Morgan, MD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Morgan PJ, Cunningham L, Mitra S, Wong N, Wu W, Noguera V, Li M, Semple J. Surgical safety checklist: implementation in an ambulatory surgical facility. Can J Anaesth. 2013 Jun;60(6):528-38. doi: 10.1007/s12630-013-9916-8. Epub 2013 Mar 16. PMID 23504355